CLINICAL TRIAL: NCT01381302
Title: Association of Polymorphism in Genes Associated With Control of Dopamine Levels in Parkinson's Disease and Tc-99m-Trodat-1 SPECT Imaging.
Brief Title: Trodat 1 SPECT and Dopamine Polymorphism
Status: Completed | Type: Observational
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Mordechai Lorberboym Prof, pI, Wolfson Medical Center
Other Study IDs: 0033-11-WOMC
Record Dates: First submitted 2011-06-14; First posted 2011-06-27 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Parkinson Disease
Keywords: Severity of disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples with DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parkinson: Early onset of disease

SUMMARY:
The study population will include 100 parkinsonian patients in early stage of disease, with total duration not exeeding 5 years.

The patients will undergo neurologic examination and evaluation of disease severity using the unified PD rating scale. Subsequently a brain SPECT will be performed using Tc-99m-Trodat1.

DETAILED DESCRIPTION:
The study sample will include 100 Israeli Jewish patients with early idiopathic PD who were not treated with anti-parkinson drugs. The clinical diagnosis will be based on the criteria of the United Kingdom Parkinson Disease Society Brain Bank.5 All patients will undergo Tc-99m-Trodat1 SPECT. The severity of the motor symptoms will be assessed with the Unified PD Rating Scale (UPDRS). Genomic DNA is extracted from peripheral blood leukocytes for genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were

1. early Israeli PD patients
2. Of jewish origin, males or females
3. Undergoing DAT-scan examination in Wolfson medical center at early stage of disease, accompanied by a UPDRS evaluation at that stage,performed by a trained neurologist
4. Patients did not use any type of anti-parkinsonian drug type, at time of DAT-scan performance and UPDRS evaluation
5. DNA sample was obtained
6. Patients were able to sign an informed consent form to participate in this study.

Exclusion Criteria:

* Patients were excluded if they features secondary parkinsonism or if they were treated with medications that block dopamine receptors.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 early Israeli PD patients Of jewish origin, males or females Undergoing DAT-scan examination in Wolfson medical center at early stage of disease, accompanied by a UPDRS evaluation at that stage,performed by a trained neurologist
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Disease severity versus genetic polymorphism | 1 year
  Correlation of disease severity with polymorphism and with striatal affinity to the DAT ligand.

SECONDARY OUTCOMES:
Severity of PD compared to specific striatal DAT activity as measures by Tc-99m Trodat SPECT. | 1 year
  For each striatal ROI, mean counts will be measured, and specific TRODAT uptake will be calculated, according to the following formula: Specific TRODAT uptake = (mean activity in ROI - mean Activity in occipital cortex) / mean Activity in occipital cortex).

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Lorberboym, MD, Principal Investigator — Edith Wolfson Medical Center
Locations (2):
- Israel (2):
  - Edith Wolfson Medical Center, Holon, Israel
  - Edith Wolfson medical Center, Holon